CLINICAL TRIAL: NCT04607044
Title: Lower Extremity Fixation In Neuropathic Patients Study
Acronym: FINS
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: US20-SAL-001
Record Dates: First submitted 2020-10-13; First posted 2020-10-28 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Neuropathy; Charcot; Disease (Etiology)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: SALVATION™ EXTERNAL FIXATION — Wright Medical's lower extremity devices used to treat neuropathic patients
  Other Names: SALVATION™ FUSION BOLTS AND BEAMS; SALVATION™ MIDFOOT NAIL; THE SALVATION™ 3DI PLATING SYSTEM; VALOR™ NAIL; HOFFMANN® LRF SYSTEM; T2® ICF SYSTEM

SUMMARY:
Prospective, multi-site, multi-year post-market clinical follow-up study on neuropathic patients treated/implanted with SALVATION™ External Fixation, SALVATION™ Fusion Bolts and Beams, SALVATION™ Midfoot Nail, The SALVATION™ 3Di Plating System, VALOR™ NAIL, HOFFMANN® LRF SYSTEM and/or T2® ICF SYSTEM of 200 patients with up to 10 sites

DETAILED DESCRIPTION:
The selected design is a US, multi-center, multi-year, non-randomized, prospective observational study. The study subjects included are neuropathic patients treated/implanted with SALVATION™ External Fixation, SALVATION™ Fusion Bolts and Beams, SALVATION™ Midfoot Nail, The SALVATION™ 3Di Plating System, VALOR™ NAIL, HOFFMANN® LRF SYSTEM and/or T2® ICF SYSTEM of 200 patients with up to 10 sites.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or non-pregnant female age 18 years or older at the time of surgery;
* Subject is willing and able to give written informed consent and comply with the requirements of this Clinical Investigation Plan (CIP); and
* Subject has neuropathy and is intended to be treated for deformity with the one or a combination of the below Systems in accordance with the legally cleared/ approved IFU and Surgical Technique Manual.
* HOFFMANN® LRF SYSTEM
* SALVATION™ EXTERNAL FIXATION SYSTEM
* SALVATION™ FUSION BOLTS AND BEAMS
* SALVATION™ 2 MIDFOOT NAIL
* SALVATION™ 3DI PLATING SYSTEM
* T2® ICF SYSTEM
* VALOR™ ANKLE FUSIO NAIL SYSTEM

Exclusion Criteria:

* Subjects determined, by the investigator, to be an inappropriate candidate for the procedure indicated;
* Unable to consent to participate (written, informed consent);
* Unable to attend/complete the requested follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neuropathic Patients treated/implanted with SALVATION™ External Fixation, SALVATION™ Fusion Bolts and Beams, SALVATION™ Midfoot Nail, The SALVATION™ 3Di Plating System, VALOR™ NAIL, HOFFMANN® LRF SYSTEM and/or T2® ICF SYSTEM
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma and Extremities
Locations (3):
- United States (3):
  - Florida Joint Care Institute, Trinity, Florida
  - Premier Orthopaedic and Sports Medicine, West Chester, Pennsylvania
  - Central Tennessee Foot and Ankle Center, Sparta, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Wright Medicals Lower Extremity Devices Used to Treat Neuropathic Patients: Wright Medicals Lower Extremity devices used to treat Neuropathic Patients
Period: Overall Study
Arm/Group | Wright Medicals Lower Extremity Devices Used to Treat Neuropathic Patients
Started | 45 (3 subjects did not receive a study device (prior to study early termination). 42 Subjects received at least one of the study devices.)
Completed | 0
Not Completed | 45
Not completed — Study Early Termination by Sponsor. | 40
Not completed — Adverse Event | 1
Not completed — Did not receive study device | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Wright Medicals Lower Extremity Devices Used to Treat Neuropathic Patients: SALVATION™ External Fixation, SALVATION™ Fusion Bolts and Beams, SALVATION™ Midfoot Nail, The SALVATION™ 3Di Plating System, VALOR™ NAIL, HOFFMANN® LRF SYSTEM and/or T2® ICF SYSTEM
Arm/Group | Wright Medicals Lower Extremity Devices Used to Treat Neuropathic Patients
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.09 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Survival Analysis of Implants at 1 Year
Description: Compare the pooled cumulative 3-year amputation (above or below the knee) rate of neuropathic patients implanted with SALVATION™ External Fixation, SALVATION™ Fusion Bolts and Beams, SALVATION™ Midfoot Nail, The SALVATION™ 3Di Plating System, VALOR™ NAIL, HOFFMANN® LRF SYSTEM and/or T2® ICF SYSTEM derived from a Kaplan-Meier survival analysis to a performance goal.
Time Frame: 1 years
Population: Given the early termination of the study the device failure analysis is through to 1 year as opposed to 3 years. 42 Subjects received the study device(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Wright Medicals Lower Extremity Devices Used to Treat Neuropathic Patients
Number analyzed (Participants) | 42
Participants | 1

2. Secondary Outcome: EQ-5D-5L- Index
Description: Evaluate improvements in patient-reported pain, function, and social interaction for quality of life from pre-op through each annual visit as assessed by the EQ-5D-5L and its component scores. Health state index scores generally range from less than 0 to 1 with higher scores indicating higher health utility. The health state preferences often represent national or regional values and can therefore differ between countries/regions.
Time Frame: 1 year
Population: Only 31 out of 42 subjects had data available at the 1 year time point for EQ-5D-5L Index.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Wright Medicals Lower Extremity Devices Used to Treat Neuropathic Patients
Number analyzed (Participants) | 31
score on scale | 0.88 (0.11)

3. Secondary Outcome: FAAM-ADL
Description: The FAAM has been shown to be valid and responsive in assessing diabetic foot disease and includes 2 subscales: Activities of Daily Living (ADL) Subscale (21 items) and Sports Subscale (8 items). For each subscale patients are asked to answer each question with a single response that most clearly describes their condition within the past week: no difficulty (4 points), slight difficulty (3 points), moderate difficulty (2 points), extreme difficulty (1 point), and unable to do (0 points). To calculate the score for either subscale, the total number of points are added (84 for the ADL subscale and 32 for the sports subscale) and converted to a percentage. A higher score reflects a higher level of physical function.
Time Frame: 1 years
Population: The patient did not complete the Sports subscale post-operatively due to physician instructions to avoid those types of activities, so FAAM results reflect the ADL subscore exclusively. A total of 7 out of 42 subjects had available data at the 1 year time point for FAAM-ADL.
Measure: Mean (Standard Deviation); unit: percentage of total score
Arm/Group | Wright Medicals Lower Extremity Devices Used to Treat Neuropathic Patients
Number analyzed (Participants) | 7
percentage of total score | 96.9 (2.85)

4. Secondary Outcome: Survival Analysis of Implants at 5 Years
Description: Compare the pooled cumulative 5-year amputation (above or below the knee) rate of neuropathic patients implanted with SALVATION™ External Fixation, SALVATION™ Fusion Bolts and Beams, SALVATION™ Midfoot Nail, The SALVATION™ 3Di Plating System, VALOR™ NAIL, HOFFMANN® LRF SYSTEM and/or T2® ICF SYSTEM derived from a Kaplan-Meier survival analysis to a performance goal.
Time Frame: 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Radiographic Assessment
Description: Assess fusion and consolidation time of bony unions utilizing surgeon's evaluations of standard of care x-rays
Time Frame: 5 years
Reporting Status: Not Posted

6. Secondary Outcome: EQ-5D-5L-VAS
Description: The second part of the EQ-5D-5L questionnaire consists of a visual analogue scale (VAS) on which the patient rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
Time Frame: 1 Year
Population: Only 31 out of 42 subjects had data available at the 1 year time point for EQ-5D-5L VAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wright Medicals Lower Extremity Devices Used to Treat Neuropathic Patients
Number analyzed (Participants) | 31
units on a scale | 86.3 (8.80)

ADVERSE EVENTS:
Time Frame: Safety was assessed through the incidence of device related intra-operative and post-operative adverse events/incidents (AEs) from baseline through study termination, up to 1.5 years. The study planned to follow all subjects annually post-operatively for 5 years (however, the study terminated early).
Description: Procedural and device related events will be described and collected on the AE form. It is the responsibility of the operating surgeon/s to be aware and note the adverse effects from the package insert/instructions for use by the manufacturer/sponsor.
Arm/Group | Wright Medicals Lower Extremity Devices Used to Treat Neuropathic Patients
All-Cause Mortality (participants affected / at risk) | 1/42
Serious Adverse Events (participants affected / at risk) | 8/42
Other Adverse Events (participants affected / at risk) | 2/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wright Medicals Lower Extremity Devices Used to Treat Neuropathic Patients (N=42)
Infection in foot (Infections and infestations) | 1 (1) — Infection in foot
Loosen External Fixator (Product Issues) | 1 (1) — Loosen External Fixator
Broken screw with nonunion at the navicular-cuneiform joint (Product Issues) | 1 (1) — Broken screw with nonunion at the navicular-cuneiform joint
Redness and swelling lower leg and ankle (Skin and subcutaneous tissue disorders) | 1 (1) — Redness and swelling lower leg and ankle
Infected IM Nail with nonunion of ankle fusion site (Infections and infestations) | 1 (1) — Infected IM Nail with nonunion of ankle fusion site
infected wire on external fixator (Infections and infestations) | 1 (1) — infected wire on external fixator
fractured tibia (Injury, poisoning and procedural complications) | 1 (1) — fractured tibia
Abcess/cellulitis (Infections and infestations) | 1 (1) — Abcess/cellulitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wright Medicals Lower Extremity Devices Used to Treat Neuropathic Patients (N=42)
Broken screw with nonunion at the navicular-cuneiform joint (Product Issues) | 1 (1) — Broken screw with nonunion at the navicular-cuneiform joint
Redness and swelling lower leg and ankle (Skin and subcutaneous tissue disorders) | 1 (1) — Redness and swelling lower leg and ankle

LIMITATIONS AND CAVEATS:
As the study was terminated early, outcomes and adverse events can only be reported up to the date of closure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT04607044/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT04607044/SAP_001.pdf